CLINICAL TRIAL: NCT00225433
Title: Luteal Phase Recombinant FSH vs. Follicular Phase Recombinant FSH for IVF Stimulation in the Poor Responder
Brief Title: Luteal Phase FSH in the IVF Poor Responder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 803515; RRU013
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: infertility; in vitro fertilization
MeSH Terms: conditions — Infertility | interventions — follitropin beta; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Follitropin beta
  Interventions: Drug: follitropin beta
- 2 (Active Comparator): Ganirelix acetate
  Interventions: Drug: ganirelix acetate

INTERVENTIONS:
Drug: follitropin beta — Follitropin beta
  Arms: 1
Drug: ganirelix acetate — Ganirelix acetate
  Arms: 2

SUMMARY:
In vitro fertilization (IVF) is a common procedure used to assist couples who have difficulty conceiving a pregnancy. IVF is a process where oocytes (eggs) are retrieved from a woman's ovaries and fertilized with sperm in the laboratory. In order to maximize the number of oocytes that can be retrieved, a women undergoes ovarian stimulation with recombinant follicle stimulating hormone (FSH). Typically 6-20 oocytes are retrieved, but in some cases there is a limited response to the stimulation, producing a limited number of oocytes. This is called poor ovarian response.

This study is designed to objectively compare two treatment regimens currently advocated in clinical practice, but never compared directly. The purpose is to assess ovarian response to starting treatment at the end of the preceding cycle may increase the number of developing oocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women planning to undergo IVF
2. Poor ovarian response in most-recent previous IVF cycle within the past 18 months as defined by the following criteria:

   A) <5 dominant follicles day of hCG, B) <5 oocytes retrieved, or C) cancellation of a previous IVF cycle due to poor response to ovulation stimulation.
3. Aged 20-42 (inclusive) at the time of randomization
4. Presence of both ovaries
5. Normal pap smear within past three years
6. At least 45 days after the last IVF cycle
7. Be willing and able to comply with the protocol for the duration of the study
8. Have given written informed consent, prior to any study-related procedure, not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

1. Clinically significant systemic disease
2. Current regular cigarette smoking by patient report
3. Known to be positive for Human Immunodeficiency Virus
4. Any medical condition which, in the judgment of the investigator and sponsor, may interfere with the absorption, distribution, metabolism or excretion of the medications used
5. Abnormal, undiagnosed gynecological bleeding
6. Known allergy or hypersensitivity to human gonadotropin preparations
7. Simultaneous participation in another investigational drug or device trial
8. Subject fails, in 2 separate menstrual cycle attempts, to have FSH ≤12.0 and an ultrasound exam within normal limits (per standard for IVF) at the Baseline Visit
9. For subjects randomized to the Luteal Phase Regimen, failure to ovulate in 2 separate menstrual cycle attempts, as evidenced by ovulation predictor kit, progesterone level, and /or visualization of corpus luteum cyst on an ovary by ultrasound exam at the Luteal Visit

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved for IVF | One cycle

SECONDARY OUTCOMES:
Number of follicles >10mm on day of human chorionic gonadotropin (hCG) administration; | 1 cycle
Number of days of stimulation; | 1 cycle
Estradiol level on the day of hCG administration; | 1 cycle
Clinical pregnancy rate per transfer: defined as the presence of an intrauterine sac on transvaginal ultrasound; | 1 cycle
Delivery rate per transfer; | 1 cycle
Safety (incidence of ovarian torsion, severe risk of ovarian hyperstimulation syndrome, enlarging hemorrhagic cysts, and serious adverse events) | 1 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States